CLINICAL TRIAL: NCT01228344
Title: Surveillance for the Effectiveness and Safety of Artemether-lumefantrine in Pediatric and Adult Patients With Malaria
Brief Title: Surveillance of Effectiveness/Safety of Artemether-lumefantrine in Patients With Malaria
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CCOA566A2424
Record Dates: First submitted 2010-10-19; First posted 2010-10-26 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Malaria
Keywords: Artemether-lumefantrine; demographics; malaria
MeSH Terms: conditions — Malaria | interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other

GROUPS / COHORTS (1):
- Artemether-lumefantrine
  Interventions: Other: Artemether-lumefantrine

INTERVENTIONS:
Other: Artemether-lumefantrine

SUMMARY:
The purpose of this study is to describe the pediatric and adult patients (U.S. and foreign residents) diagnosed with malaria and treated with artemether-lumefantrine with regard to their demographics, including evaluation of their malaria immune status, treatment effectiveness, prior and concomitant medication use, and the occurrence of adverse events in association with artemether-lumefantrine treatment, based on the information collected in the CDC Malaria Case Surveillance Report Form.

ELIGIBILITY:
Inclusion Criteria:

* Any male or female infant, child or adult patient diagnosed with malaria who received artemether-lumefantrine and was reported to the CDC. Malaria may be clinically suspected or confirmed (microscopically, and/or by polymerase chain reaction [PCR], and/or rapid diagnostic test [RDT]).

Exclusion Criteria:

* NA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any male or female infant, child or adult patient diagnosed with malaria who received artemether-lumefantrine and was reported to the Centers for Disease Control, Atlanta GA.
Sampling Method: Non-Probability Sample
Enrollment: 324 (Actual)
Dates: Start 2010-05-01 (Actual); Primary Completion 2015-09-30 (Actual); Study Completion 2015-09-30 (Actual)

PRIMARY OUTCOMES:
Effectiveness: Resolution of clinical signs and symptoms after artemether-lumefantrine treatment start | 4 weeks

SECONDARY OUTCOMES:
Adverse event, serious adverse event after artemether-lumefantrine treatment start | 4 weeks
Pregnancies after artemether-lumefantrine treatment start | Up to delivery

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Centers for Disease Control and Prevention,GA, Atlanta, Georgia, United States